CLINICAL TRIAL: NCT04303676
Title: Facilitating Alcohol Screening and Treatment (FAST), Colorado
Brief Title: Facilitating Alcohol Screening and Treatment (FAST)
Acronym: FAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-1348; 1R18HS027079-01 (AHRQ)
Record Dates: First submitted 2020-03-02; First posted 2020-03-11 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Alcohol Use Disorder
Keywords: Primary Health Care; Alcohol Drinking; Quality Improvement
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: This trial will investigate the superiority from an effectiveness perspective of: a) a virtual practice facilitation intervention, with a practice facilitator working with practices in virtual one-on-one or group sessions utilizing alcohol use e-learning modules to guide and focus the process and content, compared to b) a virtual practice facilitation intervention, with a practice facilitator working with practices in virtual one-on-one or group sessions without utilizing alcohol use e-learning modules.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Practice Facilitation with e-Learning (Active Comparator): A virtual practice facilitation intervention, with a practice facilitator working with practices in virtual one-on-one or group sessions utilizing alcohol use e-learning modules to guide and focus the process and content
  Interventions: Other: Virtual Practice Facilitation with e-Learning
- Virtual Practice Facilitation without e-Learning (Active Comparator): A virtual practice facilitation intervention, with a practice facilitator working with practices in virtual one-on-one or group sessions without utilizing alcohol use e-learning modules
  Interventions: Other: Virtual Practice Facilitation without e-Learning

INTERVENTIONS:
Other: Virtual Practice Facilitation with e-Learning — Virtual practice facilitation intervention using e-learning modules to guide the sessions includes:
  a. Practice Facilitator (PF) conducts 7 monthly virtual visits with each practice QI team i. Optional: PFs and practices may choose to conduct virtual facilitation in groups of up to 5 practices simultaneously b. MAT training (combination of virtual academic detailing plus online training resource) plus ongoing support to deal with questions through email and/or office hours with our project staff, experts, with additional consultation if needed with an addiction medicine specialist.
  c. Resources largely included as part of the e-learning module, but supplemented by online resource hub d. Centralized remote health information technology assistance, focused on implementation of registry functionality to track patients for population management and to report the measures required by AHRQ.
  Other Names: Virtual practice facilitation intervention using e-learning
  Arms: Virtual Practice Facilitation with e-Learning
Other: Virtual Practice Facilitation without e-Learning — Virtual practice facilitation intervention without e-learning to guide the sessions includes:
  a. Practice Facilitator (PF) conducts 7 monthly virtual visits with each practice QI team i. Optional: PFs and practices may choose to conduct virtual facilitation in groups of up to 5 practices simultaneously b. MAT training (virtual academic detailing) plus ongoing support to deal with questions through email and/or office hours with our project staff, experts, with additional consultation if needed with an addiction medicine specialist c. Online resource hub d. Centralized remote health information technology assistance, focused on implementation of registry functionality to track patients for population management and to report the measures required by AHRQ.
  Other Names: Virtual practice facilitation intervention without e-learning modules
  Arms: Virtual Practice Facilitation without e-Learning

SUMMARY:
Alcohol use is the third leading cause of death in the United States. Primary care practices need to implement new research findings that help identify and treat alcohol use disorder. This project will compare two methods of supporting small and medium size primary care practices in Colorado and surrounding states to improve their alcohol screening and treatment.

DETAILED DESCRIPTION:
Alcohol use causes an estimated 88,000 deaths yearly and is the third leading cause of mortality in the U.S. Unhealthy alcohol use, a spectrum from risky drinking to alcohol use disorder (AUD), impacts 27% of adults, with high cost to the health care system. Evidence-based guidelines exist for identification and treatment of unhealthy alcohol use, and evidence supports the effectiveness of medication-assisted therapy (MAT). Primary care is recognized as an ideal context for the implementation of screening and treatment processes. Despite the evidence, significant gaps exist in uptake into practice.

Practice facilitation has emerged as a key method for assisting practices in implementing organizational changes and improvements. However, in-person practice facilitation is time-intensive and costly, and virtual facilitation has not been as effective as in-person. E-learning modules can provide a structure for quality improvement in a clinical area. A pilot using e-learning combined with virtual practice facilitation was very successful from the perspectives of both practice facilitators and practices. We believe that virtual practice facilitation using e-learning modules to focus the content and process has great potential as a less costly and equally effective method compared to in-person facilitation.

In this "Facilitating Alcohol Screening and Treatment (FAST) Colorado" proposal, we will perform a cluster randomized trial to examine the Reach, Effectiveness, Adoption, Implementation, Maintenance (RE-AIM) and relative value of two approaches to supporting primary care practices to implement PCOR findings to improve their identification and treatment management of unhealthy alcohol use among adults, including screening, brief intervention, medication assisted therapy, and referral to treatment. This trial will investigate the superiority from an effectiveness perspective of: a) a virtual practice facilitation intervention, with a practice facilitator working with practices in virtual one-on-one or group sessions utilizing alcohol use e-learning modules to guide and focus the process and content, compared to b) a virtual practice facilitation intervention, with a practice facilitator working with practices in virtual one-on-one or group sessions without utilizing alcohol use e-learning modules. We will identify key practice characteristics and other contextual factors that impact the response of practices to the two practice interventions. We will compare the adaptability, trialability, and scalability of the two interventions in order to plan dissemination of the findings to key local, regional, and national stakeholders, including sharing ongoing lessons learned and resources with other programs supporting practice transformation.

ELIGIBILITY:
Inclusion Criteria: Individual patients are not directly enrolled in this study.

Practice inclusion criteria are: 1) family medicine or general internal medicine practices, generally with no more than 10 clinicians; 2) practices must be either independent or, if part of a larger organization, demonstrate that they do not receive significant QI support from the larger organization; and 3) practices must demonstrate commitment to participate fully in the intervention and evaluation, as carefully described and agreed to in a signed practice agreement. Practices with integrated behavioral health services will be included if the practice application indicates an overall level of implementation of SBIRT (screening brief intervention referral and treatment) and MAT (medication assisted treatment) that leaves room for improvement.

Exclusion Criteria:

Practices that report they have fully implemented SBIRT (screening brief intervention referral and treatment) and MAT (medication assisted treatment) for AUD (alcohol use disorder) will be excluded. Clinicians and staff who do not speak or read English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2020-05-26 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-04-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the proportion of eligible patients screened for unhealthy alcohol use | Baseline, then 3, 6, and 9 months from baseline
  Change from baseline in number and percent of eligible patients (18 years old or older) screened for unhealthy alcohol use. Change will be assessed at 3, 6, and 9 months from baseline.
Change from baseline in the proportion of screen positive patients who received brief counseling | Baseline, then 3, 6, and 9 months from baseline
  Change from baseline in the number and percent of patients who screened positive for alcohol use disorder who then received brief counseling intervention. Change will be assessed at 3, 6, and 9 months from baseline.
Change from baseline in the proportion of screen positive patients who received MAT | Baseline, then 3, 6, and 9 months from baseline
  Change from baseline in the number and percent of patients who screened positive for alcohol use disorder who then received medication assisted treatment (MAT) in the practice. Change will be assessed at 3, 6, and 9 months from baseline.
Change from baseline in the proportion of screen positive patients referred to specialty clinics | Baseline, then 3, 6, and 9 months from baseline
  Change from baseline in the number and percent of patients who screened positive for alcohol use disorder who are then referred to specialty clinics. Change will be assessed at 3, 6, and 9 months from baseline.
Change from baseline in the proportion of screen positive patients who received any treatment | Baseline, then 3, 6, and 9 months from baseline
  Change from baseline in the number and percent of patients who screened positive for alcohol use disorder who then receive at least one intervention. Change will be assessed at 3, 6, and 9 months from baseline.
Estimated cost of providing virtual practice transformation support | Up to 6 months
  The costs of providing virtual practice transformation support with and without e-learning will be estimated for the 6-month intervention period. Cost of providing practice transformation support includes both the realized cost of delivering the practice transformation support and the opportunity cost to the practice of the time providers and other practice staff working with practice facilitators as well as working independently on implementation activities.

SECONDARY OUTCOMES:
Change from baseline in the implementation of advanced primary care interventions | Baseline and at 6 months from baseline
  Comprehensive Primary Care Practice Monitor survey will assess practice-level implementation of the Building Blocks of High-performing Primary Care. Change will be assessed at 6 months from baseline.
Change from baseline in the use of evidence-based alcohol use disorder (AUD) guidelines | Baseline and at 6 months from baseline
  Practice-level assessment of (screening brief intervention referral and treatment) SBIRT and MAT activities, along with other activities aimed at AUD. An implementation checklist is completed in each practice. Change will be assessed at 6 months from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: W. Perry Dickinson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Aurora, Colorado, United States